CLINICAL TRIAL: NCT04265794
Title: Preventing Childhood Obesity Through Youth Empowerment: A Cluster RCT of the H2GO! Program
Brief Title: A Cluster Randomized Trial of the H2GO! Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University of Massachusetts, Worcester (Other); Massachusetts Alliance of Boys and Girls Clubs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-39841
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Childhood Obesity
Keywords: Sugar-sweetened beverage; Boys and Girls Clubs; Youth empowerment; Water consumption
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial (sites are randomized to the intervention or control condition)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 6-week community-based behavioral program consisting of 12 group-based weekly sessions (1-hour sessions twice a week) delivered by trained staff in the Boys and Girls Club setting. The intervention targets knowledge, attitudes, and skills related to sugar-sweetened beverage consumption and water consumption, with reduction in sugar-sweetened beverage consumption and increase in water consumption being the primary behavioral targets.
  Interventions: Behavioral: H2GO!
- Comparison (No Intervention): Parent-child pairs in comparison sites will receive usual care (standard Boys and Girls Club programming) during the study and the intervention upon study completion.

INTERVENTIONS:
Behavioral: H2GO! — Child participants will participate in a 6-week behavioral intervention consisting of 12 group-based weekly sessions (1-hour sessions twice a week) delivered by trained staff in the Boys and Girls Club setting. Each week consisted of a 1-hour health session and a 1-hour narrative session (delivered on separate days). Child participants will also receive reusable water bottles and a pictorial intervention booklet, which includes worksheets and parent-child take-home activities targeting attitudes, knowledge, and skills related to sugar-sweetened beverage and water consumption. Parent participants will be exposed to intervention messages (e.g., reduce SSB intake) through weekly parent-child take-home activities, child sharing of narratives produced, and a culminating open house event.
  Arms: Intervention

SUMMARY:
This proposal involves a collaboration with the Massachusetts Alliance of Boys and Girls Clubs. The goal is to evaluate the efficacy of youth empowerment intervention targeting sugar-sweetened beverage consumption on childhood obesity among youth. The 12-session 6-week intervention consists of health and narrative sessions and youth-led activities. For this cluster randomized controlled trial [RCT} at 10 sites, the investigators will recruit 45 parent-child pairs per site for a total of 450 parent-child pairs. The primary outcome is child participants' body mass index (BMI) z scores. Secondary outcomes include children's sugar-sweetened beverage intake, water intake, and youth empowerment. Change in outcomes over time among participants in the intervention sites will be compared to change in outcomes over time among participants

DETAILED DESCRIPTION:
Over one-third of children in the U.S. are overweight or obese and at risk for short-term and long-term health consequences, including diabetes, hypertension, heart disease and certain types of cancer. Substantial evidence exists on reducing sugar-sweetened beverage (SSB) consumption as a critical dietary target for childhood obesity prevention. Efficacious behavioral interventions targeting SSBs are lacking, particularly among low-income and ethnic minority early and pre-adolescent youth who have higher SSB intake and obesity risk. Youth empowerment interventions hold potential for catalyzing behavior change in childhood obesity intervention contexts and may be particularly engaging for low-income and ethnic minority youth. However, few studies of youth empowerment health interventions have utilized rigorous study designs or examined empowerment as a mediator/mechanism of change. To this gap, the research team has worked collaboratively with Boys and Girls Clubs of America (BGCs), a national system of after-school care that reaches 4 million youth annually, to develop and pilot-test a community-based youth empowerment intervention on reducing SSB intake and preventing childhood obesity. Grounded in Empowerment Theory, the intervention targets SSB consumption through health sessions that empower youth through developing their confidence and skills; narrative sessions that empower youth through cultivating critical thinking, and youth-led activities that empower youth through opportunities to produce change within their families. The resulting H2GO! intervention is designed to be delivered within BGCs by BGC staff. Building on the successful pilot study of H2GO!, the research team is now positioned to test the efficacy of the H2GO! intervention in collaboration with the BGC network in MA, which collectively serves over 160,000 children each year. Using a cluster-randomized design, a total of 10 BGC sites will be randomly assigned to the H2GO! intervention or a wait-list, usual care condition. A total of 450 parent-child pairs (N=45 parent-child pairs per site) will be enrolled. Data will be collected at baseline, 2 months, 6 months, and 12 months and include child anthropometrics, SSB and water intake, and youth empowerment. Specific aims of the proposal include: 1) test the efficacy of the H2GO! intervention on child BMI z scores using a cluster randomized controlled trial; 2) test the efficacy of the H2GO! intervention on child SSB and water intake; 3) examine youth empowerment as a mediator of intervention effects. Findings from this proposal will provide evidence of youth empowerment as an approach to reduce SSB intake and obesity risk and contribute to a long-term goal of producing an intervention model for childhood obesity prevention that is well-positioned for dissemination through youth-based settings.

ELIGIBILITY:
Child participant inclusion criteria

1. Ages 9-12 years
2. Current member at a BGC study site
3. Able to understand and communicate in English
4. Able and willing to provide assent
5. Parental/caregiver permission to participate

Child participant exclusion criteria - Has a medical condition that limits ability to change beverage consumption behaviors

Parent participant inclusion criteria

1. Parent or caregiver to a child member at a BGC study site
2. 18 years or older
3. able to understand and communicate in English
4. able and willing to provide consent
5. no plans to change their child's BGC membership over the next 12 months

Parent participant exclusion criteria

- has a medical condition that limits ability to change beverage consumption behaviors

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 824 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in child body mass index (BMI) z score | baseline, 12 months
  Trained staff will obtain child participants' height (inches) and weight (pounds) using standardized equipment. Height and weight will then be used to calculate BMI (kg/m^2) and BMI z scores.

SECONDARY OUTCOMES:
Change in sugar-sweetened beverage intake | Baseline, 12 months
  Sugar-sweetened beverage intake will be assessed by the self-report Beverage Intake Questionnaire (BEV-Q). Participants will report the type and quantity of sugar-sweetened beverages they consumed over the past day
Change in water intake | Baseline,12 months
  Water intake will be assessed by the self-report Beverage Intake Questionnaire (BEV-Q). Participants will report the quantity of water they consumed over the past day.

OTHER OUTCOMES:
Change in youth empowerment | Baseline,12 months
  8-item survey that asks youth to report their confidence in a range of situations using a 10-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Monica Wang, ScD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang ML, Sprague Martinez LS, Weinberg J, Alatorre S, Lemon SC, Rosal MC. A youth empowerment intervention to prevent childhood obesity: design and methods for a cluster randomized trial of the H2GO! program. BMC Public Health. 2021 Sep 15;21(1):1675. doi: 10.1186/s12889-021-11660-5. PMID 34525990